CLINICAL TRIAL: NCT06945029
Title: A Comparative Study Between Laryseal Pro Extraglottic Device and Ambu Aura Gain Laryngeal Mask as a Conduit for Fiberoptic Tracheal Intubation in Pediatric Population: A Prospective Randomized Controlled Study
Brief Title: A Comparative Study Between Laryseal Pro Extraglottic Device and Ambu Aura Gain Laryngeal Mask as a Conduit for Fiberoptic Tracheal Intubation in Pediatric Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Yahia El Sayed Kamel, Lecturer of Anesthesia, Surgical intensive care and pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: MD-38-2025
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Laryseal Pro and Ambu Aura Gain as Conduits for Fiberoptic Endotracheal Intubation

STUDY DESIGN:
Intervention Model Description: A prospective Randomized Controlled Study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambu Aura Gain extraglottic device group (Active Comparator): In this group, Ambu Aura Gain extraglottic device will be used as a conduit for fiberoptic endotracheal intubation.
  Interventions: Device: Ambu Aura Gain
- Laryseal pro extraglottic device groupI (Active Comparator): In this group, Laryseal pro extraglottic device will be used as a conduit for fiberoptic endotracheal intubation.
  Interventions: Device: Laryseal Pro

INTERVENTIONS:
Device: Ambu Aura Gain — compare between Laryseal Pro and Ambu Aura Gain extraglottic devices as conduits for fiberoptic endotracheal intubation regarding time of endotracheal intubation in pediatric population.
  Arms: Ambu Aura Gain extraglottic device group
Device: Laryseal Pro — compare between Laryseal Pro and Ambu Aura Gain extraglottic devices as conduits for fiberoptic endotracheal intubation regarding time of endotracheal intubation in pediatric
  Arms: Laryseal pro extraglottic device groupI

SUMMARY:
This study aims to compare between Laryseal Pro and Ambu Aura Gain extraglottic devices as conduits for fiberoptic endotracheal intubation regarding time of endotracheal intubation in pediatric population.

DETAILED DESCRIPTION:
Airway management is a skill that must be mastered by all anesthesiologists. Since the introduction of the extraglottic airway devices (EADs) in the early 1980s, the EAD has become a central element in the management of airway in adults and children. Some of the EADs are specially designed to allow endotracheal intubation whether blindly or with the use of fiberoptic bronchoscope (FOB). So, with the use of EAD, it is possible to provide adequate oxygenation and at the same time perform fibreoptic bronchoscopy-guided trans-device intubation, providing less hemodynamic stress response and less postoperative complications. As patient's safety always comes first, the use of flexible bronchoscopes became more widespread, strong literature favored visualization of the glottis over blind intubation. So, the use of the intubating EADs as aconduit for fiberoptic intubation is favoured over blind intubation. In addition, FOB guided intubation through EAD is a central step in the algorithm of the expected as well as the unexpected difficult airway in children.

The Ambu Aura Gain is a second-generation EAD which was presented in the clinical field in 2018. It is characterized by a wide inner diameter tunnel which has a C shaped curve with an angle guiding the endotracheal tube (ETT) into the laryngeal inlet. The presence of gastric access through a second port helps to vent the stomach and for gastric suctioning. In a previous study The Ambu Aura Gain has been shown to be an effective conduit for FOB guided intubation regarding feasibility of FOB-guided intubation, oropharyngeal leak pressure, gastric leak pressure and fibreoptic view in small children.

Laryseal Pro is a novel device and a new generation of EADs that was developed in 2018. It is believed to be a method for rapid, secure airway management which improves patient safety with gastric access. It has a catheter channel for efficient removal of fluids and gastric content, reducing risk of aspiration and integrated fenestrated flap that protects from blockage with minimal increase in flow resistance. Besides, it elevates the epiglottis for easy trauma-free ETT or bronchoscope insertion. In spite of that, it's clinical performance and efficacy as a conduit for fiberoptic tracheal intubation in pediatric population hasn't been studied by any study in literature till the present time.

To our knowledge, this is the first study to evaluate the clinical efficacy of laryseal Pro EGA in pediatric population. In this study we will compare between two extra glottic devices, Laryseal Pro and Ambu Aura Gain regarding clinical performance and efficacy with respect to the time of endotracheal intubation through fibreoptic, laryngeal view grade, airway seal pressure, success rate of intubation, number of attempts of intubation, number of attempts of SGA insertion and complications in pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Age starting from 4 years to 8 years.
* Both genders.
* ASA physical status class I-ll.
* Apparently anatomically normal with normal percentile growth chart, not suspected to have difficult airway.
* Scheduled for day case surgeries more than one hour under general anesthesia.

Exclusion Criteria:

* Parents refusal.
* Abnormality in head and neck or craniofacial anomalies as Piere Robbin syndrome, facial trauma, head and neck tumours, swellings and hemangiomas.
* Patients at risk of regurgitation and pulmonary aspiration such as patients with hiatus hernia, GERD or DM.
* Abnormal or contraindicated cervical spine flexion/extension/rotation.
* Allergy to any EAD components.
* Any active respiratory or cardiac disease and metabolic disorders.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The FOB-guided intubation time using the EAD in seconds | First 10 seconds of intubation
  the time elapsing between circuit disconnection from the EAD for the purpose of bronchoscope-guided intubation till reconnecting the circuits to the ETT and appearance of capnography waves.

CONTACTS AND LOCATIONS:
Overall Officials: Jehan A El-kholy, Professor, Study Chair — Cairo University; Maha M.I Youssef, Assistant Professor, Study Director — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No